CLINICAL TRIAL: NCT00825227
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of Armodafinil Treatment (150 mg/Day) for Patients With Fatigue Associated With Taxane Chemotherapy Alone or in Combination With Other Agents
Brief Title: Safety and Efficacy of Armodafinil for Fatigue Associated With Taxanes Alone or in Combination With Other Agents
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C10953/2036/ON/US
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Fatigue; Chemotherapy Side Effects
Keywords: Cancer; Fatigue; Taxanes
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient responses to 150 mg/day armodafinil (Active Comparator): * 150 mg/day armodafinil
  * taxane chemotherapy treatment alone or in combination with other agents
  Interventions: Drug: Armodafinil 150 mg/day
- Patient responses to placebo (Placebo Comparator): * placebo
  * taxane chemotherapy treatment alone or in combination with other agents
  Interventions: Drug: Placebo,

INTERVENTIONS:
Drug: Armodafinil 150 mg/day — * 150 mg/day armodafinil
  * concurrent with one cycle of taxane chemotherapy alone or in combination with other agents
  * patients may then continue receiving armodafinil treatment after the double-blind treatment period by entering a 24-week open-label extension period, with continuing taxane chemotherapy alone, or in combination with other agents
  Arms: Patient responses to 150 mg/day armodafinil
Drug: Placebo, — * placebo
  * concurrent with one cycle of taxane chemotherapy alone or in combination with other agents
  * patients may then continue receiving armodafinil treatment after the double-blind treatment period by entering a 24-week open-label extension period, with continuing taxane chemotherapy alone, or in combination with other agents
  Arms: Patient responses to placebo

SUMMARY:
Evaluate the Safety and Efficacy of Armodafinil Treatment for Patients With Fatigue Associated With Taxane Chemotherapy Alone or in Combination With Other Agents

DETAILED DESCRIPTION:
The primary objective of study was to determine whether armodafinil treatment at a dose of 150 mg/day is more effective than placebo treatment in reducing fatigue in patients receiving taxane chemotherapy alone or in combination with other agents by comparing the change from Screening cycle to treatment cycle (cycle 2) in the patient's average daily rating of their worst fatigue severity during the past 24 hours. In addition, the change in the percentage of days with severe fatigue and the mean Brief Fatigue Inventory scores were to be recorded.

ELIGIBILITY:
Key Inclusion Criteria:

* The patient has cancer and is receiving, or is scheduled to receive, taxane chemotherapy (paclitaxel, docetaxel, or albumin-bound paclitaxel), either alone or in combination with other agents.
* The patient experiences an average score of 6 or greater for the daily worst fatigue severity assessment during screening.
* The patient has a life expectancy of at least 6 months.
* The patient is able to use the wrist actigraphy device or provide written documentation during the screening period.
* The patient has stable hemoglobin (≥10 g/dL) throughout the screening period.
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception (including abstinence) and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
* Men not surgically sterile or who are capable of producing offspring must practice abstinence or use a barrier method of birth control, and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
* The patient has adequate hepatic and renal function.
* The patient meets the proposed diagnostic criteria for cancer-related fatigue as included in the International Classifications of Disease, Tenth Revision, Clinical Modification (ICD-10-CM).
* If the patient is taking any other chronic medication which may affect fatigue (e.g., antidepressants, anxiolytics, opioid analgesics), the dose has been stable for at least 4 weeks prior to screening and is expected to remain stable during the study.

Key Exclusion Criteria:

* The patient has any untreated reversible medical condition which may cause fatigue (e.g., metabolic disturbance, infection, endocrine abnormalities).
* The patient has received concurrent stimulant medication (e.g., dextroamphetamine or methylphenidate) during the screening period or double-blind treatment period.
* The patient has received concurrent modafinil during the screening period or double-blind treatment period.
* The patient has any delay in chemotherapy treatment such that the screening period extends beyond 6 weeks.
* The patient has known central nervous system (CNS) involvement by metastatic cancer.
* The patient is receiving concurrent radiation therapy (except for palliative radiation) or treatment with another investigational agent.
* The patient has any serious, uncontrolled, non-malignant medical or psychiatric disorder that could impair the conduct of the study or the safety of the patient.
* The patient is pregnant or lactating.
* The patient has known HIV positivity.
* The patient has nausea and vomiting or any gastrointestinal disorder that is severe enough to interfere with study drug absorption in the opinion of the investigator.
* The patient has uncontrolled pain.
* The patient has a known hypersensitivity to the study medication or ingredients of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (29):
- United States (29):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Saint Joseph Medical Center, Burbank, California
  - Compassionate Cancer Center, Fountain Valley, California
  - Wilshire Oncology, La Verne, California
  - Compassionate Cancer Center, Riverside, California
  - Scripps Cancer Center, San Diego, California
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Southeastern Gynecologic Oncology, LLC, Atlanta, Georgia
  - Augusta Oncology, Augusta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Summit Cancer Center, Savannah, Georgia
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Iowa Blood and Cancer Care PLC, Cedar Rapids, Iowa
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - Montana Cancer Institute, Missoula, Montana
  - Sparta Cancer Center, Sparta, New Jersey
  - Forsyth Regional Cancer Center, Winton, North Carolina
  - Cancer Care Associates, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Charleston Hematology Oncology, PA, Charleston, South Carolina
  - C. Michael Jones, Germantown, Tennessee
  - McLeod Cancer and Blood Center, Johnson City, Tennessee
  - Cancer Outreach Assoc. / Outreach Clinical Trial Consortium, Abingdon, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- 150 mg/Day Armodafinil: * 150 mg/day armodafinil
  * taxane chemotherapy treatment alone or in combination with other agents
- Matching Placebo: * placebo
  * taxane chemotherapy treatment alone or in combination with other agents
Period: Overall Study
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (3.73) | 56.5 (5.80) | 58.3 (4.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change Over Time in the Patient's Daily Ratings of Their Worst Fatigue Severity (as Assessed for the Past 24 Hours), Obtained From the Patient's Responses on the Brief Fatigue Inventory (BFI) Questionnaire
Description: Brief Fatigue Inventory (BFI) measures fatigue severity and impact on function on 11-point scale (0-10). Primary outcome measure is average daily rating of BFI question 3: worst level of fatigue over past 24-hours. 0 = no fatigue, 10 = worst imaginable. Study was terminated after only a few patients enrolled and therefore efficacy results were not analyzed and are not reported. Maximum response (most fatigue) would score 10 and minimum response (least fatigue) would score 0. Change was measured from Baseline (cycle 1) to cycle 2. Changes based on matching baseline period with cycle 2 period.
Time Frame: Recorded once daily by the Patient, for up to 8 weeks total (Screening and Double-Blind)
Population: Study was discontinued after only 6 subjects were enrolled due to a business decision, so no outcome analysis was done.
Groups:
- Placebo: * Placebo (3 tablets matching armodafinil tablets)
  * taxane chemotherapy treatment alone or in combination with other agents
- Armodafinil 150 mg/Day: * 150 mg/day armodafinil (3 tablets of 50 mg armodafinil)
  * taxane chemotherapy treatment alone or in combination with other agents
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Days With Severe Fatigue, From Patient Responses to the Brief Fatigue Inventory (BFI) Assessment Questionnaire
Description: The Brief Fatigue Inventory (BFI) measures severity of fatigue and impact of fatigue on daily functioning in past 24 hours. It is a 9-item questionnaire that uses an 11-point scale (0-10) to assess severity. 0 represents no fatigue, 10 represents as bad as you can imagine. The percentage of days with severe fatigue as assessed by the BFI was to be assessed. Study was terminated as a result of a business decision after only a few patients were enrolled and therefore efficacy results were not analyzed and are not reported.
Time Frame: Duration of up to 8 weeks total (Screening and Double-Blind)
Population: This trial was discontinued early after only 10 of 160 planned subjects had been recruited. No efficacy data was analyzed.
Groups:
- Patient Responses to 150 mg/Day Armodafinil: * 150 mg/day armodafinil
  * taxane chemotherapy treatment alone or in combination with other agents
  Armodafinil 150 mg/day: - 150 mg/day armodafinil
  * concurrent with one cycle of taxane chemotherapy alone or in combination with other agents
  * patients may then continue receiving armodafinil treatment after the double-blind treatment period by entering a 24-week open-label extension period, with continuing taxane chemotherapy alone, or in combination with other agents
- Patient Responses to Placebo: * placebo
  * taxane chemotherapy treatment alone or in combination with other agents
  Placebo,: - placebo
  * concurrent with one cycle of taxane chemotherapy alone or in combination with other agents
  * patients may then continue receiving armodafinil treatment after the double-blind treatment period by entering a 24-week open-label extension period, with continuing taxane chemotherapy alone, or in combination with other agents
Arm/Group | Patient Responses to 150 mg/Day Armodafinil | Patient Responses to Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in the Brief Fatigue Inventory (BFI) Global Score
Description: The Brief Fatigue Inventory (BFI) measures severity of fatigue and impact of fatigue on daily functioning in past 24 hours. It is a 9-item questionnaire that uses an 11-point scale (0-10) to assess severity. Question 3 asks for worst level of fatigue during past 24-hours. 0 represents no fatigue, 10 represents as bad as you can imagine. The global score (0 to 90) determined by adding each item was to be assessed. Study was terminated as a result of a business decision after only a few patients were enrolled and therefore efficacy results were not analyzed and are not reported.
Time Frame: Duration of up to 8 weeks total (Screening and Double-Blind)
Population: as for outcome 2
Arm/Group | Patient Responses to 150 mg/Day Armodafinil | Patient Responses to Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study drug was administered during cycle 2 of taxane therapy which lasted 21 or 28 days. This was followed by a 24-week open-label extension period during which they received armodafinil for a total of 28 weeks during which adverse events were collected.
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/4
Other Adverse Events (participants affected / at risk) | 5/6 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 mg/Day Armodafinil (N=6) | Matching Placebo (N=4)
Disease Progression (Prostate Cancer) / Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 150 mg/Day Armodafinil (N=6) | Matching Placebo (N=4)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Skin turgor decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This trial was discontinued early after only 10 of 160 planned subjects had been recruited. No efficacy data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days